CLINICAL TRIAL: NCT04764266
Title: Glycocalyx Damage During Normothermic Graft Perfusion in Orthotopic Liver Transplantation - A Pilot Study
Brief Title: Glycocalyx During Normothermic Machine Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Glycocalyx during NMP
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2022-04

CONDITIONS: Glycocalyx; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normothermic Machine Perfusion (Experimental): Blood sampling at 5 time points after transplantation Perfusate collection at 3 time points during normothermic machine perfusion prior to transplantation
  Interventions: Diagnostic Test: Heparansulfate and Syndecan 1

INTERVENTIONS:
Diagnostic Test: Heparansulfate and Syndecan 1 — Blood samples will be collected from the patient at 5 different time points. Three perfusate samples will be collected during normothermic machine perfusion (4,9ml each).

SUMMARY:
An organ intended for transplantation is normally stored on ice (cold storage, CS) after explantation from the donor. During this storage process, damage to the endothelial glycocalyx occurs. It is known from numerous studies that the integrity of the endothelial glycocalyx is necessary for organ function. Normothermic machine perfusion is an alternative storage method for explanted livers, where the graft is perfused with warm blood. This study aims to clarify the influence of normothermic machine perfusion on endothelial glycocalyx damage of the graft.

ELIGIBILITY:
Inclusion Criteria:

* First deceased donor liver transplantation receiving a graft after normothermic machine perfusion
* Recipient age >18 years
* Written informed consent

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Syndecan 1 level during normothermic machine perfusion | 24 hours
  Syndecan 1 level at the end of normothermic perfusion compared to the beginning of perfusion
Heparansulfate level during normothermic machine perfusion | 24 hours
  Heparansulfate level at the end of normothermic perfusion compared to the beginning of perfusion

SECONDARY OUTCOMES:
Syndecan 1 after transplantation | 72 hours
  Change of Syndecan 1 level after transplantation
Heparansulfate level after transplantation | 72 hours
  Change of Syndecan 1 level after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mathis, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Department of Anesthesia and Intensive Care Medicine, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No